CLINICAL TRIAL: NCT04910724
Title: Effects of Varying Energy Deficits on Protein Turnover at Rest and Carbohydrate Oxidation During Steady-state Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21-09HC
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Energy Supply; Deficiency, Severe; Energy Supply; Deficiency; Stress, Physiological

STUDY DESIGN:
Intervention Model Description: Randomized, parallel study comparing the effects of 3 magnitudes of energy deficit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 20% Energy Deficit (Experimental): Energy Deficit equal to 20% total daily energy requirements.
  Interventions: Other: Energy Deficit
- 40% Energy Deficit (Experimental): Energy Deficit equal to 40% total daily energy requirements.
  Interventions: Other: Energy Deficit
- 60% Energy Deficit (Experimental): Energy Deficit equal to 60% total daily energy requirements.
  Interventions: Other: Energy Deficit

INTERVENTIONS:
Other: Energy Deficit — A combination of individualized exercise performed on a cycle ergometer and individualized dietary prescriptions will be used to achieve energy balance or the assigned energy deficits throughout the controlled feeding and testing periods

SUMMARY:
This randomized, parallel study will examine the effects of energy balance and varying magnitudes of energy deficit on 1) the protein kinetic responses to consuming high quality protein and 2) carbohydrate oxidation during steady-state exercise. Healthy adults, representative of active duty military personnel, will complete a 2 d energy balance phase followed by a randomly assigned, 5 d energy deficit phase (n=15 per group; 20%, 40% and 60% energy deficit). At the end of each energy phase the effects of energy balance and energy deficit severity on resting postabsorptive (fasting) and postprandial (after consuming ~34 g protein) muscle protein synthesis (MPS) and whole-body protein synthesis, breakdown, and balance (synthesis - breakdown) will be determined. On the next day, the effects energy balance and energy deficit severity on carbohydrate oxidation during steady-state exercise will be determined. Primary study procedures include anthropometric and body composition measures, resting metabolic rate measures, aerobic exercise, tightly controlled diet and exercise interventions, repeated blood sampling, stable isotope infusion, stable isotope ingestion, and percutaneous muscle biopsies. The following hypotheses will be tested: 1) Δ (postprandial - postabsorptive) MPS and Δ whole-body protein balance at rest will progressively decrease as magnitude of energy deficit increases and 2) exogenous carbohydrate oxidation will be higher and endogenous carbohydrate oxidation will be lower during steady-state exercise as magnitude of energy deficit increases.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 35 years
* Body mass index < 30.0 kg/m2
* Weight stable for the past 2 months (± ~2.27 kg)
* Healthy without evidence of chronic illness or musculoskeletal injury as determined by the US Army Research Institute of Environmental Medicine Office of Medical Support and Oversight (OMSO) or home duty station medical support
* Routinely participate in aerobic and/or resistance exercise at least 2 days per week defined by self-report for previous 6 months
* Willing to refrain from taking any nonsteroidal anti-inflammatory drugs (e.g., aspirin, Advil®, Aleve®, Naprosyn®), or any other aspirin-containing product for 10 days before the first muscle biopsy and at least 5 days after completing the last muscle biopsy
* Willing to refrain from alcohol, smoking/using any nicotine product (includes e-cigarettes, vaping, chewing tobacco), caffeine, and dietary supplements during the intervention periods of the study
* Supervisor approval for federal civilian employees and non-Natick Soldier Systems Center Human Research Volunteer (HRV) active duty military personnel
* Females must have normal menstrual cycles between 26-32 days in duration; 5 menstrual cycles within the past 6 months; or able to provide documentation of oral/hormonal contraceptive use which contains low-dose estrogen/progesterone to maintain continuous levels throughout the 28-day cycle (i.e., no placebos)

Exclusion Criteria:

* Metabolic or cardiovascular abnormalities, gastrointestinal disorders (e.g., kidney disease, diabetes, cardiovascular disease, etc.)
* Significantly abnormal blood clotting as determined by OMSO or home duty station medical support
* History of complications with lidocaine
* Present condition of alcoholism, anabolic steroid use, or other substance abuse issues as determined by OMSO or home duty station medical support
* Blood donation within 8-wk of beginning the study
* Pregnant, trying to become pregnant, and/or breastfeeding (results of urine pregnancy test and self-report for breastfeeding will be obtained before body composition testing)
* Unwilling or unable to consume study diets or foods provided due to personal preference, dietary restrictions, and/or food allergies
* Unwilling or unable to adhere to study physical restrictions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Whole-body protein balance | 2 days
  Determined using L-[1-13C]-leucine stable isotope.
Muscle Protein Synthesis | 2 days
  Determined using L-[ring-2H5]-phenylalanine stable isotope.
Carbohydrate Oxidation during Steady-state Exercise | 2 days
  Determined using U-13C-glucose stable isotope.

CONTACTS AND LOCATIONS:
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT04910724/ICF_000.pdf